CLINICAL TRIAL: NCT07232511
Title: Differences in Exercise-induced Hypoalgesia After a Session With Different Blood Flow Restriction Protocols in People With Rotator Cuff-related Shoulder Pain
Brief Title: Exercise-induced Hypoalgesia Effects of Blood Flow Restriction in People With Rotator Cuff-related Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Adrián Escriche Escuder, PhD, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-FIS-3945738
Record Dates: First submitted 2025-09-26; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Related Shoulder Pain
Keywords: blood flow restriction; exercise; rotator cuff-related shoulder pain
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Resistance exercise with low blood occlusion (Experimental): A single session of exercise, 30% repetition maximum, and 30% blood occlusion
  Interventions: Device: Resistance exercise with low AOP
- Resistance exercise with moderate blood occlusion (Experimental): A single session of exercise, 30% repetition maximum, and 50% blood occlusion
  Interventions: Device: Resistance exercise with moderate BFR
- Resistance exercise with high blood occlusion (Experimental): A single session of exercise, 30% repetition maximum, and 70% blood occlusion
  Interventions: Device: Resistance exercise with high BFR
- Resistance exercise with sham blood flow restriction (Sham Comparator): A single session of exercise, 30% repetition maximum, and without blood restriction (cuff applied without pressure)
  Interventions: Device: Resistance exercise with sham BFR

INTERVENTIONS:
Device: Resistance exercise with low AOP — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 30% RM and a 30% of arterial occlusion pressure. 30" rest between sets, 2' rest between exercises.
  Arms: Resistance exercise with low blood occlusion
Device: Resistance exercise with moderate BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 30% RM and a 50% of arterial occlusion pressure. 30" rest between sets, 2' rest between exercises.
  Arms: Resistance exercise with moderate blood occlusion
Device: Resistance exercise with high BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 30% RM and a 70% of arterial occlusion pressure. 30" rest between sets, 2' rest between exercises.
  Arms: Resistance exercise with high blood occlusion
Device: Resistance exercise with sham BFR — Three exercises: external rotation at 0°, internal rotation at 0° and elevation in the scapular plane. 4 sets (30, 15, 15, reps to fatigue) with a intensity of 30% RM and a sham blood flow restriction application (cuff applied without pressure). 30" rest between sets, 2' rest between exercises.
  Arms: Resistance exercise with sham blood flow restriction

SUMMARY:
This study aims to compare the effects of blood flow restricted (BFR) exercise and to examine the differences between various BFR protocols on acute pain reduction in individuals with rotator cuff-related shoulder pain, as well as the exercise tolerance at each intensity and occlusion setting. There are four exercise modalities corresponding to different combinations of intensity (%RM) and percentage of occlusion (%AOP): 1) 30% RM and 30% AOP; 2) 30% RM and 50% AOP; 3) 30% RM and 70% AOP; 4) 30% RM and BFR placebo (cuff without pressure).

All participants will complete one session of each of the four exercise modalities, analyzing the variables studied in each for subsequent analysis and comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65
* Shoulder symptoms lasting at least 3 months
* Pain in the proximal anterolateral aspect of the shoulder, aggravated by abduction
* At least two of the following tests positive: Jobe test, resisted external rotation test, Hawkins-Kennedy test, Neer test, painful arc between 60 and 120 degrees of shoulder abduction

Exclusion Criteria:

* History of shoulder trauma or surgery
* Pain of such intensity that it is impossible to perform the proposed exercises
* Active arm elevation less than 90 degrees
* Clinical signs of a complete tear (positive delayed external and internal rotation sign and positive arm drop test)
* Suspected frozen shoulder (50% reduction or more than 30° loss in passive shoulder external rotation)
* Primary diagnosis of shoulder instability or acromioclavicular pathology
* Shoulder pain due to primary involvement in the cervical or thoracic region
* Corticosteroid injections in the last 6 weeks
* Presence of diseases such as inflammatory arthritis, neurological diseases, fibromyalgia, malignant tumors, or polymyalgia rheumatica
* Presence of more than one risk factor for thromboembolism
* Participation in upper limb exercise programs in the last month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity at rest (Visual Analogue Scale, 0-10) | Periprocedural
  Pain intensity perceived on a Visual Analogue Scale, at rest, being 0 no pain and 10 the worst pain imaginable.
Pain intensity during movement (Visual Analogue Scale, 0-10) | Periprocedural
  Pain intensity perceived on a Visual Analogue Scale during movement (flexion and abduction movement without load), being 0 no pain and 10 the worst pain imaginable

SECONDARY OUTCOMES:
Pressure pain threshold | Periprocedural
  Pressure pain threshold measured in the middle deltoid (peripheral sensitivity) and tibialis anterior (central sensitivity), using an algometer
Exercise tolerance with each setting | Periprocedural
  Exercise tolerance with each setting according to the following 5-point scale: well tolerated, tolerated, neutral, poorly tolerated, not tolerated.
Occurrence of adverse effects | Immediately after the intervention, 1 hour, 6 hours, 24 hours
  Occurrence of adverse effects (e.g., pain, delayed onset muscle soreness, sudden weakness of the trained limb, redness or swelling of the trained limb, etc.) by self-report.
Surface electromyography | Periprocedural
  Surface electromyography for the study of muscle recruitment (middle deltoid, infraspinatus, teres minor and trapezius muscles)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Escriche-Escuder, PhD, Principal Investigator — University of Valencia

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study will be available from the corresponding author upon reasonable request.